CLINICAL TRIAL: NCT04870879
Title: Colorectal Metastasis and Liver Transplantation With Organs From Deceased Donors: an Inductive Padova Center Protocol
Brief Title: Colorectal Metastasis and Liver Transplantation With Organs From Deceased Donors
Acronym: MELODIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Prof, Azienda Ospedaliera di Padova
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOP1840
Record Dates: First submitted 2021-02-23; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Liver Metastases; Colorectal Adenocarcinoma; Unresectable Malignant Neoplasm
MeSH Terms: interventions — Liver Transplantation; Drug Therapy

STUDY DESIGN:
Intervention Model Description: The study will compared survival in patient enrolled in the MELODIC trial with the OS in a matched cohort of patients treated with chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Experimental): Liver transplant
  Interventions: Procedure: Liver Transplant
- Parallel arm (Other): Chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: Liver Transplant — Liver Transplant from cadaveric donors
  Arms: Study arm
Drug: Chemotherapy — Chemotherapy
  Arms: Parallel arm

SUMMARY:
MELODIC trial is an prospective, multicenter, non-randomized, open-label, parallel trial, aimed at assessing the efficacy (in terms of overall survival: OS) of liver transplantation (LT) in unresecable CRC liver-only metastases, compared with a matched cohort of patients bearing the same tumor characteristics, and treated with chemotherapy. Synthesis of Inclusion parameters: "10;10;10;100"

ELIGIBILITY:
Inclusion Criteria (Sythesis: 10;10;10;100):

* ≥ 18 and <70 years
* Performance status, ECOG 0-1
* Histologically proved adenocarcinoma in colon or rectum.
* BRAF wild-type CRC on primary tumor or liver metastases
* High standard oncological surgical resection of the primary tumor
* Liver metastases not eligible for curative liver resection confirmed by the validation committee
* At least one line (3 months) of chemotherapy
* No signs of extra hepatic metastatic disease or local recurrence on CT, MRI and Pet-CT within 4 weeks prior to the faculty meeting at the transplant unit
* Before start of chemotherapy no lesion should be larger than > 10 cm
* Objective response according to RECIST 1.1 or SD at two consecutive CT without CEA increase
* Patient with less than 10% response on chemotherapy may be included if they obtain al least 20% response after TACE (DEB-IRI) or by 90Y-spheres
* At least 10 months time span from CRC resection and date of being listed on the transplantation list.
* Satisfactory blood tests Hb >10g/dL, neutrophils >1.0, Bilirubin<2 x upper normal level, AST, ALT<5 x upper normal level, creatinine and albumin in normal level.
* CEA<100 ng/ml
* Signed informed consent and expected cooperation of the patients for the treatment and follow up

Exclusion Criteria:

* Weight loss >10% the last 6 months
* Patient BMI > 30
* Participation refusal
* General contraindication to LT
* Prior extra hepatic metastatic disease or primary tumor local relapse.
* Other malignancies in the previous 5 years
* Pregnancy or breast feeding
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
Overall survival | 5 years

SECONDARY OUTCOMES:
Progression free survival | 3 and 5 years
Proportion of drop out | within liver transplant
Complication rate | 90 days after liver transplant

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Cillo, MD, Principal Investigator — U.O.C Chirurgia Epatobiliare e dei Trapianti Epatici, AOPD
Locations (1):
- U.O.C Chirurgia Epatobiliare e Trapianti Epatici, Azienda Ospedaliera di Padova, Padua, Italy